CLINICAL TRIAL: NCT00025051
Title: A Phase II, Double-Blind, Placebo-Controlled Clinical Trial To Assess Celecoxib As A Chemopreventive Agent Inhibiting UV-Induced Erythema And Cutaneous Carcinogenesis As Assessed Through Surrogate Biological Markers In Biopsied Skin After Exposure Of Skin In Normal Volunteers Ages 20-60 Years Old With Fitzpatrick Type I, II, III And IV Skin To UV-Radiation From Artificial Light Sources
Brief Title: Celecoxib in Preventing Skin Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000068840; CPMC-U19-CA81888-01-UV; CPMC-IRB-9923; NCI-P01-0191
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2006-12

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Celecoxib; Biological Therapy; Chemoprevention

INTERVENTIONS:
Drug: celecoxib
Procedure: anti-cytokine therapy
Procedure: antiangiogenesis therapy
Procedure: biological therapy
Procedure: cancer prevention intervention
Procedure: chemoprevention of cancer
Procedure: growth factor antagonist therapy

SUMMARY:
RATIONALE: Celecoxib may be effective in preventing skin cancer by decreasing redness caused by exposure to ultraviolet light and changing potential skin cancer biomarkers. It is not yet known whether celecoxib is more effective than a placebo in preventing skin cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of celecoxib in preventing skin cancer in participants exposed to ultraviolet light.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether celecoxib decreases ultraviolet(UV)-induced erythema and affects surrogate biomarkers of potential neoplastic change in participants with Fitzpatrick type I-IV skin exposed to UV light.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Participants are randomized to one of two treatment arms.

* Arm I: Participants receive oral celecoxib twice daily for approximately 120 days.
* Arm II: Participants receive oral placebo twice daily for approximately 120 days.

Skin biopsies of UV-exposed sites are evaluated.

Participants are followed for up to 5 weeks post-treatment.

PROJECTED ACCRUAL: A total of 36 participants (18 per arm) will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Fitzpatrick type I-IV skin
* No history of photosensitivity (e.g., systemic or discoid lupus erythematosus, polymorphous light eruption, or photocontact dermatitis)
* No history of abnormal tanning responses or other unusual reactions to natural or artificial light sources
* Willing to wear sun-protective clothing and SPF 15-49 sunscreen
* Willing and able to restrict the frequency of high ultraviolet-exposure activities (e.g., exposure to sunlight, tanning boxes, or other artificial light sources)
* No history of keloid formation

PATIENT CHARACTERISTICS:

Age:

* 20 to 60

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC ≥ 3,500/mm^3
* Hemoglobin ≥ 12.0 g/dL
* No bleeding disorder

Hepatic:

* Bilirubin ≤ 20% above upper limit of normal (ULN)
* AST and ALT ≤ 20% above ULN
* No chronic or acute hepatic disease

Renal:

* Creatinine ≤ 20% above ULN
* No chronic or acute renal disease

Gastrointestinal:

* No active gastrointestinal disease (e.g., inflammatory bowel disease)
* No pancreatic disease
* No esophageal, gastric, pyloric channel, or duodenal ulceration

Other:

* No invasive cancer except nonmelanoma skin cancer cured by excision or stage I cervical cancer
* No hypersensitivity or adverse reactions to NSAIDs, salicylates, cyclo-oxygenase-2 (COX-2) inhibitors, or sulfonamides
* No condition that would preclude the use of NSAIDs
* No clinically significant laboratory abnormalities
* No medical or psychosocial condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent chemo-immunotherapy

Chemotherapy:

* See Biologic therapy
* At least 1 year since prior chemotherapy, including topical fluorouracil

Endocrine therapy:

* At least 2 weeks since prior topical glucocorticoids
* At least 30 days since prior systemic corticosteroids
* No concurrent systemic glucocorticoids (inhaled corticosteroids allowed)
* No concurrent topical corticosteroids
* No concurrent hormonal therapy
* Hormone replacement (e.g., estrogen or thyroid replacement) allowed

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 14 days since prior aspirin (> 100 mg/day) or other non-steroidal anti-inflammatory drugs (NSAIDs) taken at least 3 times per week
* At least 2 weeks since prior topical alpha hydroxy acids (e.g., glycolic acid or lactic acid)
* At least 6 months since prior oral retinoids (3 months for topical retinoids to the face)
* At least 30 days since prior treatment for esophageal, gastric, pyloric channel, or duodenal ulceration
* At least 30 days since prior investigational medication
* No other concurrent investigational medication
* No concurrent topical vitamin A derivatives and/or alpha hydroxy acids
* No concurrent immunosuppressive drugs
* No concurrent topical medication to the skin, including prescription and over-the-counter preparations (moisturizers and emollients allowed)
* No concurrent lithium, fluconazole, or warfarin
* No concurrent chronic NSAIDs (> 3 times per week for > 2 consecutive weeks per year)
* Concurrent cardioprotective doses of aspirin (≤ 100 mg/day) allowed
* Concurrent acetaminophen allowed
* No concurrent green tea consumption of > 2 cups per day

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Bickers, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States